CLINICAL TRIAL: NCT04893733
Title: The Use of Intravenous Vitamin B Complex Improves Renal Recovery in Patients With Acute Kidney Injury
Brief Title: Intravenous Administration of Vitamin B Complex Improves Renal Recovery in Patients With AKI
Acronym: VIBAKI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Caja Nacional de Salud (Other)
Collaborators: International Society of Nephrology (Other)
Responsible Party: Principal Investigator, Rolando Claure-Del Granado, MD, Head Division of Nephrology, Caja Nacional de Salud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBCNS
Record Dates: First submitted 2021-05-16; First posted 2021-05-19 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2022-07

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Vitamin B complex; Creatinine; Proteinuria
MeSH Terms: conditions — Acute Kidney Injury; Proteinuria | interventions — Vitamin B Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin B complex (Experimental): Randomized patients with AKI to this arm will received during 5 consecutive days IV Vitamin B complex each 12 hours.
  Interventions: Drug: Vitamin B Complex; Other: STOP AKI protocol

INTERVENTIONS:
Drug: Vitamin B Complex — Patients with established AKI will be randomized to received IV vitamin B complex each 1 hours for 5 consecutive days versus placebo.
  Every patients will also received Institution standard of care for AKI
  Other Names: Complejo B Vimin
Other: STOP AKI protocol — STOP AKI protocols includes:
  S: identify and treat sepsis. Standard measures should be followed to decrease the risk of infection. Close surveillance to identify early signs of infection with appropriate treatment T: avoid nephrotoxins. Avoidance of drugs harmful to the kidneys (e.g. NSAIDs, gentamicin) Care with intravenous iodinated contrast O: optimize blood pressure and optimize volume status. Avoid dehydration e.g. confused patient. Treat hypovolaemia promptly. Consider with-holding patient anti-hypertensives/diuretics until assessed after major surgery or if patient develops sepsis/hypovolemia P: Prevent harm. Identify the cause promptly and manage appropriately to prevent progression. Prevent complications by instituting prompt therapy. Identify drugs excreted through the kidneys and adjust drug doses promptly if AKI develops. Review fluid management plans to prevent inadequate or excessive intravenous fluid administration

SUMMARY:
Animal and human studies have shown that the administration of vitamin B3 (niacin) improves renal ischemia; helping to recover from acute kidney injury (AKI) more effectively; Therefore, its use in patients with AKI could improve short-term outcomes: accelerating the recovery of renal function, reducing the days of hospital stay and costs; as well as reducing the incidence of chronic kidney disease (CKD) or progression of CKD after an episode of AKI.

Our main objective is to determine the usefulness of the administration of vitamin B complex as a treatment for established acute kidney injury and its effect on short and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who meet modified KDIGO criteria for Acute Kidney Injury, based on serum creatinine or urinary volume criteria.

Exclusion Criteria:

* Patient under 18 years of age
* Patients with stage G5 chronic kidney disease
* Patients with chronic kidney replacement therapy.
* Pregnant women
* Transplant patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Complete renal recovery | Day 7
  Serum creatinine (CrS) level returns to its baseline value or to a lower value.

SECONDARY OUTCOMES:
Progression to Acute Kidney Disease (AKD) | 1 month
  A eGFR < than 60 ml/m/1.73m2
De novo chronic kidney disease (CKD) | 3 months
  An eGFR < than 60 ml/m/1.73m2
Progression of CKD | 3 months
  Patients progresses from a lower KDIGO CKD stage to a higher CKD stage

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Claure-Del Granado, M.D., Principal Investigator — Hospital Obrero No 2 - C.N.S.
Locations (1):
- Hospital Obrero No 2 - C.N.S., Cochabamba, Departamento de Cochabamba, Bolivia

IPD SHARING:
Plan to Share IPD: No